CLINICAL TRIAL: NCT06033703
Title: Topical Netarsudil for the Prevention of Proliferative Vitreoretinopathy in Patients With Primary Rhegmatogenous Detachments and Retinal Detachment Due to Proliferative Vitreoretinopathy or Open-Globe Injury: A Phase I/II Clinical Trial
Brief Title: Topical Netarsudil for the Prevention of Proliferative Vitreoretinopathy in Patients With Retinal Detachment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Leo Am Kim, M.D., Assistant Professor of Ophthalmology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022P000152
Record Dates: First submitted 2023-08-17; First posted 2023-09-13 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Rhegmatogenous Retinal Detachment; Proliferative Vitreoretinopathy
Keywords: Vitrectomy; Netarsudil; Pharmacokinetics; Safety; Efficacy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Primary retinal detachment, Phakic group (Experimental): Phakic patients with primary rhegmatogenous retinal detachment repair within 7 days of symptom onset, undergoing vitrectomy or vitrectomy with scleral buckle will be included.
  Patients will receive topical Netarsudil ophthalmic solution 0.02%: once per day, from time of diagnosis of retinal detachment to 16 weeks post-operatively.
  Interventions: Drug: Netarsudil Ophthalmic
- Primary retinal detachment, Pseudophakic group (Experimental): Pseudophakic patients with primary rhegmatogenous retinal detachment repair within 7 days of symptom onset, undergoing vitrectomy or vitrectomy with scleral buckle will be included.
  Patients will receive topical Netarsudil ophthalmic solution 0.02%: once per day, from time of diagnosis of retinal detachment to 16 weeks post-operatively.
  Interventions: Drug: Netarsudil Ophthalmic
- Secondary retinal detachment, Phakic group (Experimental): Phakic patients with retinal detachment due with proliferative vitreoretinopathy (grade C or higher) or retinal detachment associated with open globe trauma, undergoing vitrectomy or vitrectomy with scleral buckle will be included.
  Patients will receive topical Netarsudil ophthalmic solution 0.02%: once per day, from time of diagnosis of retinal detachment to 16 weeks post-operatively.
  Interventions: Drug: Netarsudil Ophthalmic
- Secondary retinal detachment, Pseudophakic group (Experimental): Pseudophakic patients with retinal detachment due with proliferative vitreoretinopathy (grade C or higher) or retinal detachment associated with open globe trauma, undergoing vitrectomy or vitrectomy with scleral buckle will be included.
  Patients will receive topical Netarsudil ophthalmic solution 0.02%: once per day, from time of diagnosis of retinal detachment to 16 weeks post-operatively.
  Interventions: Drug: Netarsudil Ophthalmic

INTERVENTIONS:
Drug: Netarsudil Ophthalmic — Topical administration of Netarsudil
  Other Names: Rhopressa

SUMMARY:
This study has two main objectives. The first objective is to study the pharmacokinetics of topical netarsudil administration in the posterior segment of the eye, where netarsudil must exert its effect in order to prevent formation of tractional membranes.

The second objective is to assess the safety profile of topical netarsudil in the pre- and post-operative periods. A secondary objective of the study is to begin to assess signs of efficacy in preventing formation of tractional membranes post-operatively.

DETAILED DESCRIPTION:
This is an open-label, randomized study that will test the safety and pharmacokinetics of topical netarsudil at a dose frequency of once-daily in two cohorts of patients: those with primary rhegmatogenous detachments, and those with established proliferative vitreoretinopathy. The intervention will be topical application of Netarsudil from time of diagnosis of retinal detachment to 16 weeks post-operatively.

Patients will be randomized to one of the following groups:

* The primary rhegmatogenous detachment cohort: A total of 24 study subjects (24 eyes) will be stratified by their lens status (12 phakic versus 12 pseudophakic). All patients will receive once per day dosing of netarsudil.
* The proliferative vitreoretinopathy cohort: A total of 24 study subjects (24 eyes) will be stratified by their lens status (12 phakic versus 12 pseudophakic). All patients will receive once per day dosing of netarsudil.

After surgery, patients will continue on once per day dosing of Netarsudil for a total of 16 weeks post-op.

ELIGIBILITY:
The primary rhegmatogenous detachment cohort will have the following selection criteria:

Inclusion criteria:

* Patients > 18 years old
* Patients presenting for primary rhegmatogenous retinal detachment repair within 28 days of symptom onset
* Patients undergoing vitrectomy or vitrectomy with scleral buckle

Exclusion criteria:

* Patient unable to give consent
* Patient unable to follow-up
* Prior history of retinal detachment incisional surgery in presenting eye
* Prior history of open globe injury to presenting eye
* Prior history of glaucoma surgery to presenting eye I.e., Status post trabeculectomy, Ahmed tube placement, minimally invasive glaucoma surgery, actively on glaucoma medication
* Prior history of corneal disease, or history of corneal edema
* Patient already on topical netarsudil in presenting eye
* Patient without natural lens or intraocular lens implant (I.e., aphakic patients)
* Patients with intraocular pressure <8mm Hg in operative eye
* Active or chronic or recurrent uncontrolled ocular or systemic disease
* Active or history of chronic or recurrent inflammatory eye disease
* Diagnosis of proliferative diabetic retinopathy
* Signs of ocular infection at presentation in either eye
* Known or suspected sensitivity or allergy to any of the medications used in the operation or postoperatively
* Inability to use/ apply topical eye drops

The proliferative vitreoretinopathy cohort will have the following selection criteria:

Inclusion criteria:

* Patients > 18 years old
* Patient presenting with retinal detachment due with proliferative vitreoretinopathy (grade C or higher) or retinal detachment associated with open globe trauma
* Patients undergoing vitrectomy or vitrectomy with scleral buckle

Exclusion criteria:

* Patient unable to give consent
* Patient unable to follow-up
* Prior history of glaucoma surgery to presenting eye I.e., Status post trabeculectomy, Ahmed tube placement, minimally invasive glaucoma surgery
* Patient already on topical netarsudil in presenting eye
* Patients with intraocular pressure <8mm Hg in operative eye
* Active or chronic or recurrent uncontrolled ocular or systemic disease
* Active or history of chronic or recurrent inflammatory eye disease
* Diagnosis of severe nonproliferative or proliferative diabetic retinopathy or vasoproliferative disease in operative eye
* Signs of ocular infection at presentation in either eye
* Known or suspected sensitivity or allergy to any of the medications used in the operation or postoperatively
* Inability to use/ apply topical eye drops
* No Light Perception vision in operative eye
* Failure to achieve intraoperative reattachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The concentration of netarsudil in the vitreous to assess its pharmacokinetic properties. | Through study completion, an average of 1 year
  Netarsudil concentration in the posterior segment of the eye, using High-performance liquid chromatography (HPLC)
Serious adverse events | Day 1, 7, 28, 84, and 168 after surgery
  Unexpected serious adverse events

SECONDARY OUTCOMES:
Number of operations within 3 months | Day 84 after surgery
  Total number of operation during the first 3 months after surgery
Final attachment status at last follow-up | Day 168 after surgery
  Status of the retina (attached versus detached) at last follow-up visit
Visual acuity | Day 1, 7, 28, 84, and 168 after surgery
  Best-corrected visual acuity measured using Snellen chart
Spectral domain optical coherence tomography (SD-OCT) of the macula | Day 1, 7, 28, 84, and 168 after surgery
  Status of the macula (mac-on versus mac-off)
Adverse events | Day 1, 7, 28, 84, and 168 after surgery
  Adverse events including conjunctival injection, subconjunctival hemorrhage, and corneal verticillata, eye irritation, reticular edema of the cornea, hypotony

CONTACTS AND LOCATIONS:
Overall Officials: Leo Kim, MD, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Mass Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CW, Sherman B, Moore LA, Laethem CL, Lu DW, Pattabiraman PP, Rao PV, deLong MA, Kopczynski CC. Discovery and Preclinical Development of Netarsudil, a Novel Ocular Hypotensive Agent for the Treatment of Glaucoma. J Ocul Pharmacol Ther. 2018 Jan/Feb;34(1-2):40-51. doi: 10.1089/jop.2017.0023. Epub 2017 Jun 13. PMID 28609185
- [Background] Singh IP, Fechtner RD, Myers JS, Kim T, Usner DW, McKee H, Sheng H, Lewis RA, Heah T, Kopczynski CC. Pooled Efficacy and Safety Profile of Netarsudil Ophthalmic Solution 0.02% in Patients With Open-angle Glaucoma or Ocular Hypertension. J Glaucoma. 2020 Oct;29(10):878-884. doi: 10.1097/IJG.0000000000001634. PMID 32826769
- [Background] Davies E, Jurkunas U, Pineda R 2nd. Pilot Study of Corneal Clearance With the Use of a Rho-Kinase Inhibitor After Descemetorhexis Without Endothelial Keratoplasty for Fuchs Endothelial Corneal Dystrophy. Cornea. 2021 Jul 1;40(7):899-902. doi: 10.1097/ICO.0000000000002691. PMID 33758139
- [Background] Kahook MY, Serle JB, Mah FS, Kim T, Raizman MB, Heah T, Ramirez-Davis N, Kopczynski CC, Usner DW, Novack GD; ROCKET-2 Study Group. Long-term Safety and Ocular Hypotensive Efficacy Evaluation of Netarsudil Ophthalmic Solution: Rho Kinase Elevated IOP Treatment Trial (ROCKET-2). Am J Ophthalmol. 2019 Apr;200:130-137. doi: 10.1016/j.ajo.2019.01.003. Epub 2019 Jan 15. PMID 30653957
- [Background] Serle JB, Katz LJ, McLaurin E, Heah T, Ramirez-Davis N, Usner DW, Novack GD, Kopczynski CC; ROCKET-1 and ROCKET-2 Study Groups. Two Phase 3 Clinical Trials Comparing the Safety and Efficacy of Netarsudil to Timolol in Patients With Elevated Intraocular Pressure: Rho Kinase Elevated IOP Treatment Trial 1 and 2 (ROCKET-1 and ROCKET-2). Am J Ophthalmol. 2018 Feb;186:116-127. doi: 10.1016/j.ajo.2017.11.019. Epub 2017 Dec 1. PMID 29199013
- [Background] Fernandez MM. Reticular Epithelial Edema in Edematous Corneas Treated with Netarsudil. Ophthalmology. 2018 Nov;125(11):1709. doi: 10.1016/j.ophtha.2018.08.004. No abstract available. PMID 30318038
- [Background] Wisely CE, Liu KC, Gupta D, Carlson AN, Asrani SG, Kim T. Reticular Bullous Epithelial Edema in Corneas Treated with Netarsudil: A Case Series. Am J Ophthalmol. 2020 Sep;217:20-26. doi: 10.1016/j.ajo.2020.04.002. Epub 2020 Apr 11. PMID 32289295
- [Background] LoBue SA, Moustafa GA, Vu A, Amin M, Nguyen T, Goyal H. Transient Reticular Cystic Corneal Epithelial Edema With Topical Netarsudil: A Case Series and Review. Cornea. 2021 Aug 1;40(8):1048-1054. doi: 10.1097/ICO.0000000000002621. PMID 33369939